CLINICAL TRIAL: NCT05199155
Title: Phase II Study Evaluating the Safety and Efficacy of NerVFIX Treatment for Trauma or Accidental Nerve Section of the Wrist
Brief Title: Use of a Nerve Regeneration Conduit (NerVFIX®) in the Treatment of Nerve Section of the Wrist
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: TBF Genie Tissulaire (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NerVFIX-TBF2; 2019-A03050-57 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-12-30; First posted 2022-01-20 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Nerve Injury; Nerve Lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NerVFIX (Experimental): Biological regeneration nerve conduit of allogeneic artery or vein from umbilical cord used as a conduit for gap < 2 cm or as a wrap after peripheral nerve suture
  Interventions: Biological: NerVFIX

INTERVENTIONS:
Biological: NerVFIX — Decellularized, freeze-dried and sterile allogeneic graft of artery or vein from umbilical cord use by the investigator as a nerve regeneration conduit

SUMMARY:
The purpose of this open, multicenter trial is to assess the impact of a nerve regeneration conduit made of allogeneic artery or vein from umbilical cord lining on the regeneration of wrist nerve.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age and under 65 years of age
* One wrist nerve section ( medial, ulnar) with a minimum of 2 mm and maximum gap of 2 cm evaluated during the surgical procedure (Sunderland Grade V)
* Inclusion of direct suture with wrapping or nerve defect with NerVFIX for nerve junction
* Poor outcome on the Mackinnon-Dellon scale: < S3
* Within 1 month of the injury or accident event and/or at the time of the injury (emergency procedure)
* Any damaged artery must be repaired
* Patient with no poor vascularization risk (no surgical treatment of vessel section) or no disease linked to poor vascularization.
* Patient who received the study information and provided consent
* Patients who are members or the beneficiary of a national health insurance plan

Exclusion Criteria:

* Breast feeding women or women without effective contraception (if no effective contraception: a pregnancy test is mandatory)
* Digital nerve section
* Pregnant or breast feeding women: Women of childbearing age will be asked to undergo a pregnancy test before being enrolled into the study and to use an effective birth control method
* Patient who suffered amputation of the hand in question
* Surgical site infection or necrotic area; tendon and/or bone damage
* Underlying motor or sensory disorder that could compromise the evaluation; inflammatory arthritis causing pain
* Disease that compromises healing such as diabetes, alcoholism or skin disorder
* Vascular disease leading to reduced blood flow or altered microvascularisation such as Raynaud's disease
* Subjects who are unlikely to follow through with rehabilitation or who could be addicted to drugs or alcohol; heavy smokers will be asked to stop smoking voluntarily
* Persons confined by a judicial or administrative decision
* Adults subject to legal protection measures or who are unable to provide their consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Recovery of sensory function | 12 months
  Recovery of sensitivity in the nerve section area evaluated using the static 2-Point Discrimination (s2PD)

SECONDARY OUTCOMES:
Progressive recovery of sensory function | 15 days, 1 month, 3 months, 6 months, 12 months
  Improvement in the s2PD
Decrease of the score of symptoms related to nerve section | 15 days, 1 month, 3 months, 6 months, 12 months
  Score of cold sensitivity, hyperaesthesia and numbing (0 = no complication, 4 = major complication) and score of pain to the pressure (0 = no pain, 10 = worst imaginable pain)
Improvement of the touch-pressure threshold of the hand | 15 days, 1 month, 3 months, 6 months, 12 months
  Touch-pressure of the hand in grammes determined using Semmes-Weinstein Monofilament (SWM) tests
Percentage of nerve regeneration | 1 month, 3 months, 6 months, 12 months
  Nerve regeneration after surgical repair evaluated by Hoffman-Tinel sign
Improvement of health-related quality of life | 15 days, 1 month, 3 months, 6 months, 12 months
  Quality of life related to nerve section of the hand evaluated using Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire (0 = no disability, 100 = most severe disability)
Improvement of clinical motricity | 15 days, 1 month, 3 months, 6 months, 12 months
  Improvement of thumb opposition in case of median nerve section or of Froment's sign, abduction and adduction of the fingers and movement of the 4th and 5th digit in case of ulnar nerve section

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique de la Main - Nantes Atlantique, Saint-Herblain
  - Institut Chirurgical de la Main et du Membre Supérieur, Villeurbanne

IPD SHARING:
Plan to Share IPD: No